CLINICAL TRIAL: NCT03123523
Title: Study of the Relation Between Lipid Myocardial Overload Evaluated by Cardiac Magnetic Resonance Imaging (MRI), Alteration of Longitudinal Myocardial Deformations by Echocardiography, and Clinical Achievements (Functional, Biological and Electrical) in Fabry Disease, and Its Outcomes.
Acronym: FABRY-Image
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/08
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — Exercise Test; Biological Assay

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients group: 35 patients
  Interventions: Diagnostic Test: Echocardiography at T0; Diagnostic Test: Exercise test; Biological: Biological assays; Device: MRI with contrast agent injection; Diagnostic Test: Echocardiography at M24
- Healthy volunteers: 20 healthy volunteers
  Interventions: Diagnostic Test: Echocardiography at T0; Device: MRI without contrast agent injection

INTERVENTIONS:
Diagnostic Test: Echocardiography at T0
Diagnostic Test: Exercise test
  Groups: Patients group
Biological: Biological assays — Creatinin, hematocrit and BNP assays
  Groups: Patients group
Device: MRI with contrast agent injection — With injection of gadolinium
  Groups: Patients group
Device: MRI without contrast agent injection — Without injection of gadolinium
  Groups: Healthy volunteers
Diagnostic Test: Echocardiography at M24
  Groups: Patients group

SUMMARY:
Anderson-Fabry disease is a genetic lysosomal storage disease, linked to chromosome X (gene GLA), responsible of enzyme synthesis deficit in α-galactosidase A with intracellular sphingolipids accumulation and multiorganic achievement.

If renal complication is principally responsible of the pejorative evolution of the disease, it may also exist a cardiac achievement, symptomatic or not (heart failure symptoms including dyspnea, conduction abnormalities, supra-ventricular and ventricular arrhythmias), with or without left ventricular hypertrophy (LVH).

Administration of agalsidase-α or ß, a genetic engineering synthetic equivalent of the deficient enzyme, should significantly slow disease evolution indeed reduce LVH.

Some patients with Fabry disease without LVH should present, compared to healthy subjects, indirect early markers of intramyocyte lipid overload:

* in echocardiography, longitudinal myocardial deformation (strain) should be altered while ejection fraction is preserved, and
* in cardiac MRI, T1 mapping should be reduced1. This was also previously demonstrated in Fabry patients with LVH2. However, are these abnormalities of longitudinal deformation in echocardiography and of T1 mapping in MRI correlated to the presence of pejorative cardiac markers (such as clinical and functional tolerances, Brain Natriuretic Peptide (BNP) level and electrical complications)?

ELIGIBILITY:
Inclusion Criteria:

Patients group :

* Adults (age ≥18 years), male and female.
* Patients diagnosed genetically having Fabry disease, with or without clinical cardiac symptoms and with different evolution stades of the disease.
* For female in age of procreation, efficient contraception will be required and a negative pregnancy test.
* Oral agreement of the patient after having read information note.
* Patient affiliated to social national Security registry.

Healthy volunteers group:

* Adults (age ≥18 years), male and female.
* Unscathed of cardiovascular pathologies and cardiovascular risk factors.
* For female in age of procreation, efficient contraception will be required and a negative pregnancy test.
* Oral agreement of the patient after having read information note.
* Patient affiliated to social national Security registry.

Exclusion Criteria:

For the 2 groups :

* Extracardiac pathology limiting life expectancy <1 year (cancer).
* Pregnant or breastfeeding female.
* Claustrophobia.
* Mechanical prosthetic valve.
* Severe obesity > 140 kg
* Patients with intracardiac device (implantable cardiac defibrillator, pace maker, resynchronisation), surgical clips not MRI compatible, neurosensorial stimulators, cochlear implants, ferromagnetic foreign bodies (ocular, cerebral), neurosurgical derivation valves)
* Impossibility to provide consent or refusal to sign the consent form.

For the patients:

- Previous history of hypersensitivity to gadolinium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - The 35 patients will be selected from Dr Réant (Cardiologist) and Dr Rooryck-Thambo's (Genetician) consultations, co-responsible of the Regional Competence Centre in Inherited Cardiomyopathies (Bordeaux, france) and from a medical specialized group following regularly these patients (Dr Valérie de Précigout in Nephrology at Bordeaux Pellegrin Hospital, Pr Cyril Goizet and Pr Didier Lacombe in Genetics at Bordeaux Pellegrin Hospital).
  Inclusion will be performed according to current management and follow-up recommendations.
  - The 20 healthy volunteers will be recruited form a local database (" HSync Study " of Dr Cornolle). Their consent will be requested at inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2016-10-18 (Actual); Primary Completion 2020-04-18 (Estimated); Study Completion 2020-04-18 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular symptoms | Baseline
  Dyspnea, angor, syncope and lipothymia, palpitations, heart failure signs
Metabolic exercise test marker : poor blood pressure adaptation to exercise | Baseline
Metabolic exercise test marker: max level achieved | Baseline
Metabolic exercise test marker : percentage of theoretical maximal heart rate | Baseline
Metabolic exercise test marker : peak of Oxygen uptake (VO2) | Baseline
Metabolic exercise test marker : percentage of expected peak VO2 | Baseline
Metabolic exercise test marker : Expiratory volume / carbon dioxide production (VE/VCO2) | Baseline
Biological marker : BNP elevation | Baseline
Electrical markers at ECG and Holter ECG | Baseline
  Measure of conduction troubles; supra-ventricular and ventricular arrhythmias.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No